CLINICAL TRIAL: NCT05072483
Title: Natural History Study of CADASIL
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000413; 000413-H
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12-16

CONDITIONS: Cardiovascular Disease; Arterial Stiffness; Germline Mutation in the NOTCH 3 Gene; Pathogenesis of CADASIL; Clinical Phenotype of CADASIL
Keywords: Biospecimen Procurement; Laboratory Research Specimens; progressive chronic hypoperfusion; Stroke; progressive white matter degeneration, and debilitating dementia.
MeSH Terms: conditions — Cardiovascular Diseases; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy controls for exploratory analyses, where the measurements were not commonly performed previously in other populations, for qualitative comparison with CADASIL population
  Interventions: Device: MRI
- Subjects with CADASIL: Adult genetically-confirmed patients with a wider range of CADASIL disease duration and debility
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Research pulse sequences.

SUMMARY:
Background:

CADASIL (cerebral autosomal dominant arteriopathy with subcortical infarct and leukoencephalopathy) is a genetic disorder. It causes narrowing of the small blood vessels and can lead to strokes and dementia. Researchers want to monitor people with CADASIL over time.

Objective:

To learn more about how CADASIL affects a person s blood vessels over time.

Eligibility:

Adults ages 18 and older who have CADASIL, and healthy volunteers.

Design:

Participants will be screened with a medical record review.

Participants will have 4 study visits over 9 years. Visits will last 6 8 hours per day, for 2 4 days.

Participants will give blood and urine samples. They will have an electrocardiogram to record their heart s electrical activity. They will fill out a family tree. They will have tests that measure mental abilities like memory and attention. They may have a skin biopsy. They may have a lumbar puncture.

Participants will have an eye exam. Their pupils will be dilated. They will receive a dye via intravenous (IV) line. Pictures will be taken of their eyes.

Participants will have an imaging scan of their brain. They may receive a contrast agent via IV.

Participants blood flow and blood vessel flexibility will be measured. In one test, a probe will be pressed against the skin of the their wrist, neck, and groin. In another test, they will hold one arm still while a microscope makes videos of the blood flow through a fingernail. In another test, they will perform light exercise or other activities while wearing an elastic band around their head or probes placed on their arm or leg.

Healthy volunteers will complete some of the above tests.

DETAILED DESCRIPTION:
Study Description:

This is a disease discovery/natural history protocol. We will enroll up to 110 CADASIL subjects with the goal of 100 CADASIL subjects completing the study to perform in-depth prospective and retrospective evaluations for research purposes and up to 45 healthy control subjects with the goal of 40 completing the study for comparison.

Objectives:

Primary Objective: This study will examine the pathogenesis and progression of CADASIL through comprehensive evaluations, and molecular studies on biospecimens collected from affected individuals.

Secondary Objective: Comprehensive evaluations will be used to investigate variability of the genotype and clinical phenotype of CADASIL during the study period.

Exploratory Objective: Healthy controls may be used for comparison for some of the research testing where data on normal values is lacking. Healthy controls will not be used to establish normal range values but for qualitative comparison with CADASIL population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligibility for this study may be determined based on information collected under other NHLBI-approved protocols, outside records and patient report.

In order to be eligible to participate in this study, an individual must meet criteria 1 & 2 and either criteria 3 or 4:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 18 to 100 years (inclusive).
3. Established diagnosis of CADASIL or NOTCH3 mutations, as determined by genetic testing.
4. Healthy controls.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or nursing at time of consent.
2. Subjects who lack capacity to consent and don't have a legally authorized representative.
3. Subjects who decline to provide samples for blood and/or tissue studies.
4. Subjects who do not speak English.
5. Subjects whose scans or examinations show unexpected brain conditions (outside of CADASIL) which would interfere with interpretation of testing.
6. Subjects unable to undergo an MRI scan or subjects meeting the following criteria:

   * Subjects who have internal non-MRI compatible metals (i.e., cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or metal fragments in the eye) as these rendering an MRI unsafe
   * Subjects with ferromagnetic dental bridges or crowns (exclusion only for 7.0T)
   * Subjects unable to remain supine for the expected length of the MRI (i.e., up to 1 hour)
   * Subjects with uncontrolled head movements
   * Subjects who are claustrophobic for the expected length of the MRI (i.e., up to 1 hour) and claustrophobia cannot be controlled with anti-anxiety medication.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will follow up to 110 subjects in order to have 100 subjects with CADASIL (at least 80 new CADASIL subjects and up to 20 CADASIL subjects previously enrolled in our pilot study, if they would like to participate in this study as well) and up to 45 healthy controls with the goal of 40 healthy control subjects completing the study, withtotal accrual of 155 male and female, ages 18-100. Should anyone from the original patient cohort decide not to participate in this new study, additional patients will be recruited in order to meet our goal of having 100 CADASIL subjects enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2034-06-01 (Estimated); Study Completion 2041-06-01 (Estimated)

PRIMARY OUTCOMES:
This study will examine the pathogenesis of CADASIL through comprehensive clinical evaluations and molecular studies on biospecimens collected under this protocol from affected individuals. | 13 years
  To study the pathogenesis of CADASIL and obtain clinical evaluations and biospecimens from affected cohorts to identify underlying disease mechanism(s).

SECONDARY OUTCOMES:
Clinical evaluations will be used to investigate variability of clinical phenotype during the study period. | 20 years
  To use Clinical evaluations to investigate variability of clinical phenotype during the study period. These studies will serve as baseline evaluations for future studies on the identification of underlying disease mechanism(s) and potential therapeutic approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa A Ferrante Brenlla, Ph.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000413-H.html